CLINICAL TRIAL: NCT04114916
Title: Clinical Trial to Evaluate the Efficacy of a Nutraceutical Versus Placebo in Reducing Cardiovascular Risk in Healthy Subjects.
Brief Title: Clinical Trial to Evaluate the Reduction of Cardiovascular Risk
Acronym: NUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-0005
Record Dates: First submitted 2018-04-19; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-01

CONDITIONS: Cholesterol
MeSH Terms: interventions — Apigenin; grapefruit seed extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apigenin, luteonin, grapefruit extract and citrolive (Experimental): One capsules a day. It will be consumed at breakfast for eight weeks.
  Interventions: Dietary Supplement: Apigenin, luteonin, grapefruit extract and citrolive
- maltodextrina (Placebo Comparator): One capsules a day. It will be consumed at breakfast for eight weeks.
  Interventions: Dietary Supplement: maltodextrina

INTERVENTIONS:
Dietary Supplement: Apigenin, luteonin, grapefruit extract and citrolive — Two capsules daily at breakfast and dinner.
  Arms: Apigenin, luteonin, grapefruit extract and citrolive
Dietary Supplement: maltodextrina — Two capsules daily at breakfast and dinner.
  Arms: maltodextrina

SUMMARY:
Randomized parallel and double blind clinical trial in which it is intended to analyze the efficacy of a nutraceutical on cholesterol and endothelial function after the consumption of a product for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (men or women) between 40 and 75 years of age, of Caucasian race
* Women must be in the menopausal period.
* Present body mass index between 18.5 and 34.9 Kg / m2.
* The number of platelets in whole blood must be greater than 170 x109 / L
* Hematocrit greater than 40% for men or greater than 35% for women.
* Hemoglobin greater than 120 g / L for men or 110 g / L for women.
* Present fasting levels of LDL-serum cholesterol equal to or greater than 110mg / dL
* Present fasting values of total serum cholesterol equal or superior to 180mg / dL
* Volunteers able to understand the clinical study and willing to give written informed consent and to comply with the procedures and requirements of the study.

Exclusion Criteria:

* Thyroid dysfunction, infections, or with any type of chronic disease (for example, autoimmune, inflammatory).
* Subjects who have suffered an ischemic-vascular event during the last months
* Subjects undergoing medication and / or nutraceutical treatment for hypertension, diabetes or hyperlipidemia (eg Statins).
* Subjects under treatment with drugs that due to their narrow therapeutic margin require monitoring of their plasma levels (digoxin, acenocoumarol, warfarin, etc ...)
* Subjects under treatment that affect body weight or appetite.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Subjects who are performing or intend to perform any type of diet, hypocaloric or not, during the conduct of the study.
* Subjects who have donated a minimum of 0.5L of blood in the last month.
* Vegetarian subjects.
* Subjects, who have ingested, in the last three months, supplements of omega 3 and / or 6, (eg fish oil, evening primrose oil, krill oil, or algae oil).
* Subjects under treatment with niacin or fibrates.
* Those subjects with alcohol abuse, or with excessive alcohol consumption (> 3 glasses of wine or beer / day) will be excluded.
* Patients undergoing major surgery in the last 3 months.
* Subjects who smoke or not, but in any case who do not modify their nicotinic habits during their participation in the study.
* Participation in another clinical trial in the three months prior to the study Lack of will or inability to comply with clinical trial procedures.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
endothelial function | The measurements of endothelial function are taken with an ultrasound on two different occasions. The measurements will be made at baseline and after eight weeks of product consumption.
  Changes in the dilatation of the Humeral artery.
blood samples | Total cholesterol measurements are taken with the ILAB 600 analyzer on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product.
  Change in total cholesterol levels.
Tests | Quality of life measurements are taken on two different occasions. Measurements are made at the beginning and after eight weeks of product consumption.
  Change in physical activity with the World Physical Activity Questionnaire (GPAQ)
nutritional record | The dietary intake will be controlled by a diary in which meals will be recorded for three days and on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product.
  Volunteers record dietary intake for three days in a notebook. They will describe the amount of food they consume in grams in order to assess changes in intake during the clinical trial.
body composition | Body measurements are taken with a Tanita on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product.
  Changes in body composition were measured with a TANITA
cardiovascular risk | Cardiovascular risk measurements are taken by laboratory analysis on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product.
  Changes in systolic blood pressure (mmHg), dystolic blood pressure (mmHg) and heart rate (beats per minute).
Tests | Quality of life measurements are taken on two different occasions. Measurements are made at the beginning and after eight weeks of product consumption.
  Change in the quality of life (SF-12).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol